CLINICAL TRIAL: NCT02250053
Title: The COURAGE Trial: Colon Recurrence and Aerobic Exercise: A Feasibility Study
Brief Title: Exercise and Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 10214
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Stage II Colon Cancer; Stage III Colon Cancer
Keywords: stage II and stage III colon cancer survivors, who have completed curative treatment i.e., surgical resection and chemotherapy for their colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: exercise
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental): aerobic exercise on soluble intercellular adhesion molecules
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
Despite the success of surgery and chemotherapy among people with colon cancer, 30-50% of patients develop recurrent disease. Physical activity has emerged as a potential lifestyle intervention to reduce cancer recurrence and improve survival among people with colon cancer (CC). This pilot study aims to identify the dose-response effects of aerobic exercise on molecular and cellular pathways associated with physical activity and CC outcomes among patients with stage II and III CC.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed TNM stage II-III CC;
2. completed surgical resection and adjuvant chemotherapy (if applicable) within 1-24 months before entering the study;
3. ≤120 min/wk of self-reported moderate or vigorous intensity physical activity using the Paffenbarger physical activity questionnaire;
4. age ≥18 years;
5. written physician approval;
6. no additional surgery planned within the 6-month intervention (including colostomy reversal);
7. ability to walk unaided for 6-minutes;
8. no contraindications to exercise using the PA readiness questionnaire (PAR-Q), unless physician approves participation with specific knowledge of this contraindication.

Exclusion Criteria:

1. history of another primary invasive cancer (other than non-melanoma skin-cancer);
2. evidence of metastatic CC (i.e., TNM M1);
3. planning to receive any additional adjuvant chemotherapy;
4. pregnant or breast feeding;
5. unable to provide baseline blood sample;
6. cardiac conditions, including the following:

   1. myocardial infarction or coronary revascularization procedure within prior 3 months;
   2. uncontrolled hypertension (systolic ≥180 mmHg or diastolic ≥100 mmHg);
   3. high-risk or uncontrolled arrhythmias;
   4. clinically significant valvular disease;
   5. decompensated heart failure;
   6. known aortic aneurysm;
7. any other condition that may impede testing of the study hypothesis or make it unsafe to engage in the exercise program (determined by the investigative team).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
1. The biological efficacy of aerobic exercise on soluble intercellular adhesion molecule-1 (sICAM-1), and soluble vascular adhesion molecule-1 (sVCAM-1) prognostic biomarkers. | 2 years

SECONDARY OUTCOMES:
Exercise adherence, quantified as the percentage of total dose completed relative to the total dose prescribed during the six-month study; | 6 months
Visceral adipose tissue and anthropometric measures at baseline and six-months; | 6 months
Fasting insulin measured at baseline and six-months; | six months
Circulating tumor cells measured at baseline and six-months. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Brown JC, Compton SLE, Meyerhardt JA, Spielmann G, Yang S. The dose-response effect of aerobic exercise on inflammation in colon cancer survivors. Front Oncol. 2023 Dec 12;13:1257767. doi: 10.3389/fonc.2023.1257767. eCollection 2023. PMID 38148846